CLINICAL TRIAL: NCT01459536
Title: Rotator Cuff Function and Muscle Morphology in Older Adults With Rotator Cuff Tear
Brief Title: Assessment of Muscle Function and Size in Older Adults With Rotator Cuff Tear
Acronym: ARC
Status: Completed | Type: Observational
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Other Study IDs: 14547
Record Dates: First submitted 2011-10-21; First posted 2011-10-25 (Estimated); Last update posted 2017-11-07 (Actual); Status verified 2017-03

CONDITIONS: Rotator Cuff Tear
Keywords: Aging
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Rotator Cuff Tear-surgical
- Health Older Adult Control
- Rotator cuff tear - non surgical

SUMMARY:
Adequate upper limb function is critically important to maintenance of independence and prevention of disability in older adults. The goal of this work is to identify factors that contribute to rotator cuff rupture and improved outcomes for repair. Ultimately, the investigators seek to identify patients most at risk for rupture and to guide clinicians on optimal surgical and rehabilitation strategies. This pilot study will quantitatively characterize the morphological (muscle volume and fatty infiltration) and functional (shoulder isometric joint strength, movement when performing typical task) changes in the muscles of the rotator cuff following supraspinatus tear and surgical repair. The investigators hypothesize that patients with supraspinatus tear will have reduced muscle volume and increased fatty infiltration of rotator cuff muscles compared to their contralateral arm and age-matched controls, which will increase following surgery. The investigators further hypothesize that isometric joint strength in these individuals will be associated with muscle volume and the degree of fatty infiltration, and that older adults with a rotator cuff tear will use a restricted range of motion to accomplish functional tasks. This study emphasizes muscle function and composition with application to rehabilitation of upper limb function, which complements the theme of the Pepper Center.

ELIGIBILITY:
Inclusion Criteria:

* adults ≥ 60 years of age
* free of any medical condition that might be exacerbated by physical testing
* patients: major thickness supraspinatus tear
* control subjects: no history of significant injury or pathology in either upper limb

Exclusion Criteria:

* contraindication to undergoing MRI
* history of neuromuscular disorder, or any injury that may affect the upper limb (e.g. any history of stroke, Parkinson's, or spinal cord injury, or being confined to a wheelchair)

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: orthopaedic surgery clinic, community sample
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2011-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Shoulder strength | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Saul, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

REFERENCES:
- [Derived] Vidt ME, Santago AC 2nd, Tuohy CJ, Poehling GG, Freehill MT, Kraft RA, Marsh AP, Hegedus EJ, Miller ME, Saul KR. Assessments of Fatty Infiltration and Muscle Atrophy From a Single Magnetic Resonance Image Slice Are Not Predictive of 3-Dimensional Measurements. Arthroscopy. 2016 Jan;32(1):128-39. doi: 10.1016/j.arthro.2015.06.035. Epub 2015 Sep 29. PMID 26391648